CLINICAL TRIAL: NCT00632008
Title: A Randomised, Double-blind, Placebo-controlled Study to Determine the Efficacy of Soluble Beta-1,3/1,6-glucan in Chronic Foot Ulcers in Diabetes
Brief Title: Soluble Beta-glucan (SBG) as Treatment for Diabetic Foot Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biotec Pharmacon ASA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBG-1-12
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Diabetic Foot Ulcers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): SBG
  Interventions: Drug: Soluble beta-glucan (SBG)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Soluble beta-glucan (SBG) — Topical application of SBG to the wound, at least twice a week until complete healing or for 8 maximum weeks
  Arms: 1
Drug: Placebo comparator — Topical application of placebo to wound, at least twice a week until compleate healing or for maximum 8 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the application of soluble beta-glucan (SBG) onto diabetic foot ulcers improves the healing of the ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes mellitus
* Age ≥ 18 years
* One or more full-thickness ulcers at or below the level of the malleoli, which do not extend to tendon, joint, or bone
* The ulcer (or index ulcer, if appropriate) must have been present for at least 4 weeks prior to Day 0 but not longer than 2 years
* Ankle:brachial pressure index (ABPI) >0.7, or the presence of two palpable pulses on the affected foot
* Ulcer area >25 mm2 but <500 mm2
* Written informed consent

Exclusion Criteria:

* Pregnancy, lactation or absence of adequate contraception for women with child bearing capacity
* ABPI < 0.7
* Serum albumin < 2.0 g/dL
* Gangrene on any part of the foot with the study ulcer
* Presence of signs of clinically significant foot infection on Day 0
* Chronic renal failure with calculated GFR <30 ml/min
* Surgical procedure (other than debridement) on the foot with the study ulcer in the 28 days prior to Day 0
* HbA1c 12% or more
* Current alcohol or drug abuse
* Participation in other studies in the preceding 28 days
* An ulcer on a foot affected by acute Charcot osteoarthropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-03; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Jeffcoate, MD, PhD, Principal Investigator — Nottingham City Hospital
Locations (11):
- United Kingdom (11):
  - Belfast City Hospital, Belfast
  - Royal Blackburn Hospital, Blackburn
  - Royal Bournemouth Hospital, Bournemouth
  - Southmead Hospital, Bristol
  - NHS Greater Glasgow and Clyde Victoria, Glasgow
  - Leeds General Infirmary, Leeds
  - Leicester General Hospital, Leicester
  - North Manchester Hospital, Manchester
  - Newcastle General Hospital, Newcastle
  - Northampton General Hospital, Northampton
  - Nottingham City Hospital, Nottingham